CLINICAL TRIAL: NCT03246386
Title: Pharmacokinetics of Posaconazole Given as a Single Intravenous Dose to Obese Subjects: Dosing Obese With Noxafil® Under a Trial (DONUT)
Brief Title: Dosing Obese With Noxafil® Under a Trial (DONUT)
Acronym: DONUT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: St. Antonius Hospital (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UMCN-AKF-17.08
Record Dates: First submitted 2017-08-02; First posted 2017-08-11 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2019-12

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — posaconazole

STUDY DESIGN:
Intervention Model Description: Comparing a 2 groups of obese subjects vs 1 group of non-obese subjects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Obese subjects (Experimental): Subjects with a BMI>35 kg/m2
  Interventions: Drug: Posaconazole Injection [Noxafil] 300mg; Drug: Posaconazole Injection [Noxafil] 400mg
- Non-obese subjects (Active Comparator): Subjects with a BMI>18.5 and <25 kg/m2
  Interventions: Drug: Posaconazole Injection [Noxafil] 300mg

INTERVENTIONS:
Drug: Posaconazole Injection [Noxafil] 300mg — Single dose by intravenous infusion 300mg
Drug: Posaconazole Injection [Noxafil] 400mg — Single dose by intravenous infusion 400mg
  Arms: Obese subjects

SUMMARY:
Although posaconazole is approved for the prophylaxes and treatment of invasive fungal infections, specific dosing guidelines for posaconazole in (morbidly) obese patients are not specified. There is clear evidence indicating that heavier patients are receiving a sub-optimal dose if the current guidelines are used. Specifically in the setting of augmented prevalence of species with intermediate susceptible to posaconazole, adequate dosing is needed at start of treatment.

Therefore it seems prudent to conduct a trial in a cohort of obese patients who receive posaconazole (300mg or 400mg) and define the pharmacokinetics. These will then be compared to the pharmacokinetics in a normal-weight group receiving 300mg posaconazole.

DETAILED DESCRIPTION:
Obese patients with a BMI ≥ 35 kg/m2 undergoing endoscopic gastric bypass surgery will receive a 300 mg or 400mg dose of posaconazole. A PK curve will be determined after administration at t=0.45, 0.75, 1, 1.5, 2, 4, 8, 12, 24, and (if feasible) 48 hours post infusion. Blood samples (4 mL) on PK days will be taken to obtain at least 2.0 mL of plasma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects BMI:

   * obese groups: subject must have a BMI ≥35 kg/m2 at the time of inclusion,
   * non-obese group: subject must have a BMI ≥18.5 and < 25kg/m2 at the time of inclusion.
2. Subject is at least 18 of age on the day of screening and not older than 65 years of age on the day of dosing;
3. If a woman, is neither pregnant nor able to become pregnant and is not nursing an infant;
4. Subject is able and willing to sign the Informed Consent before screening evaluations.

   For the non-obese subjects the following additional inclusion criteria applies:
5. Subject is in good age-appropriate health condition as established by medical history, physical examination, electrocardiography, results of biochemistry, hematology and urinalysis testing within 6 weeks prior to study drug administration. Results of biochemistry, hematology and urinalysis testing should be within the laboratory's reference ranges (see Appendix A). If laboratory results are not within the reference ranges, the subject is included based on the investigator's judgment that the observed deviations are not clinically relevant. This should be clearly recorded;

Exclusion Criteria:

1. Documented history of sensitivity to medicinal products or excipients similar to those found in the posaconazole preparation;
2. History of, or known abuse of drugs, alcohol or solvents (up until a maximum of three months before study drug administration);
3. Use of medication that has known relevant interaction with study drug as determined by the investigator up to 1 weeks prior to study drug administration.
4. Donation of blood or plasma to a blood bank or in a clinical study (except a screening visit) within 4 weeks prior to study drug administration;
5. Blood transfusion within 8 weeks prior to study drug administration;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-05 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Posaconazole exposure | Through study completion (usually after 24 or 48 hours)
  The concentration-time curve of posaconazole in obese will be compared with that in non-obese subjects. Exposure is assessed by Area-Under-the-Curve from zero to 48 hours (AUC0-48h).

SECONDARY OUTCOMES:
Exposure with augemented posaconazol dose | Through study completion (usually after 24 or 48 hours)
  The concentration-time curve of posaconazole in obese receiving 400mg will be compared with that in non-obese subjects. Exposure is assessed by Area-Under-the-Curve from zero to 48 hours (AUC0-48h).

CONTACTS AND LOCATIONS:
Overall Officials: Roger Brüggemann, PhD-PharmD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - St. Antonius hospital, Nieuwegein
  - Radboudumc, Nijmegen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wasmann RE, Smit C, van Donselaar MH, van Dongen EPA, Wiezer RMJ, Verweij PE, Burger DM, Knibbe CAJ, Bruggemann RJM. Implications for IV posaconazole dosing in the era of obesity. J Antimicrob Chemother. 2020 Apr 1;75(4):1006-1013. doi: 10.1093/jac/dkz546. PMID 31971567
- See also: paper — https://pubmed.ncbi.nlm.nih.gov/31971567/